CLINICAL TRIAL: NCT05217849
Title: Multi-domain Online Therapeutic Investigation Of Neurocognition
Brief Title: Multi-domain Online Therapeutic Investigation Of Neurocognition (MOTION)
Acronym: MOTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco VA Health Care System (U.S. Federal Agency); University of California, Los Angeles (Other); United States Department of Defense (U.S. Federal Agency); CDMRP (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-33507; CDMRP - AZ160019 (Other Grant/Funding Number: Congressionally Directed Medical Research Programs Defense Health Agency Research & Development)
Record Dates: First submitted 2021-11-16; First posted 2022-02-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Mild Cognitive Impairment; Subjective Memory Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Tai Ji; Health

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to an on-line Tai Chi class, an on-line mindful movement class, or to an on-line Health and Wellness Education classes. All classes will meet twice a week for one hour for 12-weeks. The randomization sequence will be generated in advance by Dr. Chao's research team using a random number generator and will be maintained in a secure location. Individuals who collect and analyze outcome data will be blinded to group assignment.
Who Masked: Outcomes Assessor
Masking Description: The randomization sequence will be generated in advance by Dr. Chao's research team using a random number generator and will be maintained in a secure location. Individuals who collect or analyze outcome data will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Chi (Experimental): Participants will engage in 60-minute Tai Chi classes twice a week for 12 weeks. The classes will be live-streamed over the internet. Tai Chi is an ancient Chinese system of gentle physical exercise and stretching. It involves a series of movements performed in a slow, focused manner and accompanied by deep breathing.
  Interventions: Behavioral: Tai Chi
- Gentle, Mindful Movement (Experimental): Participants will engage in a gentle, mindful movement class twice a week for 12 weeks. The classes will be one hour long and will be live-streamed over the internet. The mindful movement classes will combine elements from a wide range of Eastern and Western exercise modalities, including occupational therapy, physical therapy, yoga, tai chi, Feldenkrais, Rosen Method, dance movement therapy and mindfulness meditation.
  Interventions: Behavioral: Preventing Loss of Independence through Exercise (PLIE)
- Health and Wellness Education (Active Comparator): Participants will engage in bi-weekly 60 minute sessions of Health and Wellness Education classes. The classes will be held on-line for 12 weeks.
  Interventions: Behavioral: Health and Wellness Education

INTERVENTIONS:
Behavioral: Tai Chi — Tai Chi is an ancient Chinese form of exercise/martial art that involves a series of movements performed in a slow, focused manner and accompanied by deep breathing.
  Other Names: Tai-Chi-Chih (TCC)
  Arms: Tai Chi
Behavioral: Preventing Loss of Independence through Exercise (PLIE) — PLIE is a gentle, mindful movement exercise program that integrates elements of Eastern and Western exercise modalities to develop mindful body awareness and enhance social connection.
  Other Names: gentle, mindful movement class
  Arms: Gentle, Mindful Movement
Behavioral: Health and Wellness Education — This on-line class will consist of hour-long lectures/talks about various topics related to healthy aging and wellness.
  Arms: Health and Wellness Education

SUMMARY:
The purpose of this study is to compare the effects of three on-line wellness interventions for improving physical and cognitive function and brain connectivity in adults who are at least 55 years old and are experiencing symptoms of memory and/or cognitive difficulties.

DETAILED DESCRIPTION:
The proposed study will perform a randomized, controlled trial (RCT) to compare the effects of three on-line wellness interventions for adults (age 55 years and older) who are experiencing memory and/or cognitive decline. Study participants will be randomly assigned to one of three on-line wellness interventions: (a) Tai Chi, (b) mindful movement course, or (c) health and wellness education course. All interventions will be one hour long, held on-line twice a week for 12 weeks. The co-primary outcomes are 3-month change in cognitive function (Alzheimer's Disease Assessment Scale - cognitive subscale, ADAS-cog) and functional brain connectivity within the default mode network (DMN). Secondary behavioral outcomes will include measures of specific cognitive processes (e.g., auditory memory, executive function, processing speed), physical function (e.g., mobility), anxiety, depression, fatigue, pain, sleep quality, social activities/social isolation, and quality of life. Secondary neuroimaging outcomes will include measures of functional connectivity in other intrinsic brain networks (e.g., salience, central executive, language), cerebral perfusion, and structural white matter integrity. The behavioral and imaging outcomes will be assessed at baseline and upon completion of the 12-week interventions. To assess durability of the behavioral effects of the interventions, the cognitive and behavioral outcomes will be assessed again 6 months after the completion of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 55 years
* subjective cognitive complaints, defined as self-experienced persistent decline in cognitive capacity in comparison with a previously normal status and unrelated to an acute event
* Montreal Cognitive Assessment (MoCA) score suggestive of Mild Cognitive Impairment (MCI) status (i.e., < 26)
* English language fluency
* Wireless internet connection at home
* Willingness to travel to the San Francisco VA in northern California or UCLA in southern California for in-person assessments at baseline, after the 12-week interventions, and at the 36-week follow-up
* Capacity to provide informed consent or legally authorized representative consent and participant assent.

Exclusion Criteria:

* current or past Axis I psychiatric disorders, or recent unstable medical or neurological disorders
* disabilities that prevent participation in on-line movement classes (e.g., primarily use wheel-chair, severe visual impairment that would limit ability to observe instructor's movement on screen or severe hearing impairment that would limit ability to hear instructor's directions)
* insufficient English proficiency
* limited life expectancy (i.e., enrolled in hospice, metastatic cancer)
* plan to travel for > 1 week during 12-week intervention period
* diagnosis of dementia per the DSM-5
* MoCA score suggestive of dementia (i.e., <17)
* started dementia medication (cholinesterase inhibitor or memantine) in past 3 months or plans to start dementia medication during study period
* planning to start/change any psychoactive medication during study period
* current participation in another research study
* contraindications to magnetic resonance imaging (MRI), including claustrophobia severe enough to prevent MRI examination, presence of ferrometallic objects in the body that would interfere with MRI examination and/or cause a safety risk (e.g., pacemakers, implanted stimulators, pumps)
* prior or current training in with Tai Chi, PLIE, or other mind-body practices

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) Scores | Change from baseline to 1-week post-treatment.
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale is a brief neuropsychological assessment used to assess the severity of cognitive symptoms of dementia. ADAS-cog scores range from 0-70, with higher scores (≥ 18) indicating greater cognitive impairment.
Change in Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog) Scores | Change from baseline to 6 months after treatment ends.
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale is a brief neuropsychological assessment used to assess the severity of cognitive symptoms of dementia. ADAS-cog scores range from 0-70, with higher scores (≥ 18) indicating greater cognitive impairment.
Change in Default Mode Network (DMN) functional connectivity | Change from baseline to 1-week post-treatment.
  The default mode network (DMN) is a system of connected brain areas that show increased activity when a person is not focused on what is happening around them. Instead, the DMN is especially active when a person is engaged in introspective activities (e.g., daydreaming, or contemplating the past or future). Research suggests that the DMN is disrupted in people with Mild Cognitive Impairment (MCI) and Alzheimer's disease (AD).
  Functional connectivity can be defined as the similarity between brain signals that arise from two anatomically separated brain regions. Similarity between the brain signals can be analyzed using Pearson's correlation.

SECONDARY OUTCOMES:
Change in Auditory Memory scores | Change from baseline to 1 week post-treatment.
  The stories subtest of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) will be used to assess auditory memory. Raw scores will be transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. Thus the sample mean (across all arms) is zero for each test score. The z-scores were then averaged to produce a composite scores. Higher scores are indicative of better performance.
Change in Auditory Memory scores | Change from baseline to 6 months after treatment ends.
  The stories subtest of the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) will be used to assess auditory memory. Raw scores will be transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. Thus the sample mean (across all arms) is zero for each test score. The z-scores were then averaged to produce a composite scores. Higher scores are indicative of better performance.
Change in Attention/Executive Function Cognitive Domain Scores | Change from baseline to 1-week post-treatment.
  Neuropsychological tests will included the following domains: Attention/Executive Function (Trail Making Test A and B, Stroop Interference [Golden version])
  Raw scores will be transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. Thus the sample mean (across all arms) is zero for each test score. The z-scores will be averaged to produce composite scores. Higher scores are indicative of better performance.
Change in Attention/Executive Function Cognitive Domain Scores | Change from baseline to 6 months after treatment ends.
  Neuropsychological tests will included the following domains: Attention/Executive Function (Trail Making Test A and B, Stroop Interference [Golden version])
  Raw scores will be transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. Thus the sample mean (across all arms) is zero for each test score. The z-scores will be averaged to produce composite scores. Higher scores are indicative of better performance.
Change in Verbal Fluency scores | Change from baseline to 1-week post-treatment.
  Controlled Oral Word Association test (FAS). Raw scores will be transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. Thus the sample mean (across all arms) is zero for each test score. Higher scores are indicative of better performance.
Change in Verbal Fluency scores | Change from baseline to 6 months after treatment ends.
  Controlled Oral Word Association test (FAS). Raw scores will be transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. Thus the sample mean (across all arms) is zero for each test score. Higher scores are indicative of better performance.
Change in Processing Speed Scores | Change from baseline to 1-week post-treatment.
  Processing speed will be assessed with the coding subtest of RBANS as well as the Digit Symbol Substitution Test (DSST). Raw scores will be transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. Thus the sample mean (across all arms) is zero for each test score. The z-scores will be averaged to produce composite scores. Higher scores are indicative of better performance.
Change in Processing Speed Scores | Change from baseline to 6 months after treatment ends.
  Processing speed will be assessed with the coding subtest of RBANS as well as the Digit Symbol Substitution Test (DSST). Raw scores will be transformed to z-scores (with a mean of 0 and standard deviation of 1) for each test score of interest across all participants. Thus the sample mean (across all arms) is zero for each test score. The z-scores will be averaged to produce composite scores. Higher scores are indicative of better performance.
Change in Mobility | Change from baseline to 1-week post-treatment.
  Mobility will be assessed with the Timed Up and Go (TUG) test, which assesses the time it takes participants to stand up from a chair, walk 3 meters, turn around, walk back to the chair and sit down. In addition, we will assess steady-state gait during 90 seconds of continuous over-ground walking at normal preferred speed, with and without the addition of a dual task challenge (counting backward by one or by two).
Change in Mobility | Change from baseline to 6 months after treatment ends.
  Mobility will be assessed with the Timed Up and Go (TUG) test, which assesses the time it takes participants to stand up from a chair, walk 3 meters, turn around, walk back to the chair and sit down. In addition, we will assess steady-state gait during 90 seconds of continuous over-ground walking at normal preferred speed, with and without the addition of a dual task challenge (counting backward by one or by two).
Change in Salience Network functional connectivity | Change from baseline to 1-week post-treatment.
  The Salience Network consists of a network of brain regions whose cortical hubs are the anterior cingulate and ventral anterior insular (i.e., frontoinsular) cortices. This network also includes nodes in the amygdala, hypothalamus, ventral striatum, thalamus, and specific brainstem nuclei.
Change in Language Network functional connectivity | Change from baseline to 1-week post-treatment.
  The Language Network consists of a group of left-lateralized frontal and temporal brain regions that responds to written/spoken/signed words and sentences, but not to mental arithmetic, music perception, executive function tasks, or action/gesture perception.

OTHER OUTCOMES:
Change in PROMIS-29 Health-Related Quality of Life (HRQoL) Domains | Change from baseline to 1 week post-treatment.
  The PROMIS-29 includes seven HRQoL domains: Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, and Pain). The pain domain has two subdomains (interference and intensity). Each of the 7 domains has four 5-level items (i.e., 16 decrements each). In addition to these items, pain intensity is assessed using a single 11-point numeric rating scale anchored between no pain (0) and worse imaginable pain (10), adding 10 additional decrements.
Change in PROMIS-29 Health-Related Quality of Life (HRQoL) Domains | Change from baseline to 6 months after treatment ends.
  The PROMIS-29 includes seven HRQoL domains: Physical Functioning, Anxiety, Depression, Fatigue, Sleep Disturbance, Social Functioning, and Pain). The pain domain has two subdomains (interference and intensity). Each of the 7 domains has four 5-level items (i.e., 16 decrements each). In addition to these items, pain intensity is assessed using a single 11-point numeric rating scale anchored between no pain (0) and worse imaginable pain (10), adding 10 additional decrements.
Change in measures of body awareness | Change from baseline to 1-week post-treatment.
  We will examine 3 measures of body awareness: Interoceptive attention is the ability to sustain and control attention to body sensations. Interoceptive self-regulation is the ability to regulate distress by attention to body sensations. These two measures will be assessed with MAIA-2 self-report questionnaire. We will also utilize the Body Awareness portion of the Body Experience Questionnaire to measure interoceptive attention/awareness.
Change in measures of body awareness | Change from baseline to 6 months after treatment ends.
  We will examine 3 measures of body awareness: Interoceptive attention is the ability to sustain and control attention to body sensations. Interoceptive self-regulation is the ability to regulate distress by attention to body sensations. These two measures will be assessed with MAIA-2 self-report questionnaire. We will also utilize the Body Awareness portion of the Body Experience Questionnaire to measure interoceptive attention/awareness.
Change in a measure of mindfulness | Change from baseline to 1-week post-treatment.
  Mindfulness will be assessed with the Freiburg Mindfulness Index (FMI), a valid and reliable 30-item questionnaire measuring mindfulness.
Change in a measure of mindfulness | Change from baseline to 6 months after treatment ends.
  Mindfulness will be assessed with the Freiburg Mindfulness Index (FMI), a valid and reliable 30-item questionnaire measuring mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Linda L Chao, PhD, Principal Investigator — University of California, San Francisco & SFVAHCS
Locations (1):
- VA Health Care System, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chao LL, Barnes DE, Chesney MA, Mehling WE, Lee JA, Benjamin C, Lavretsky H, Ercoli L, Siddarth P, Narr KL. Multi-domain Online Therapeutic Investigation Of Neurocognition (MOTION) - A randomized comparative-effectiveness study of two remotely delivered mind-body interventions for older adults with cognitive decline. Contemp Clin Trials. 2025 Feb;149:107811. doi: 10.1016/j.cct.2025.107811. Epub 2025 Jan 12. PMID 39809343